CLINICAL TRIAL: NCT04863729
Title: Evaluation of Asdzáán Be'eená Teen Pregnancy and Substance Use Prevention Program for Native American Youth and Their Caregiver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Children's Bureau - Administration for Children and Families (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00014736
Record Dates: First submitted 2021-04-13; First posted 2021-04-28 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Sex Behavior
Keywords: Primary prevention; Teen pregnancy prevention; Substance use prevention; Parent-child intervention
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The program consists of 11 weekly sessions conducted with girls ages 10-14 and their female caregivers. 5 of the 11 sessions will be taught to groups of 9-13 girls and their female caregivers, and 6 of the sessions will be taught to individual girl/female caregiver dyads. The choice to use a mix of group- and individual sessions is based on findings from the formative phase indicating certain topics should be taught in groups (e.g. Navajo history and reproductive health 101), and certain topics be taught in individual dyads (e.g. family values and the clan system).
  Interventions: Behavioral: Asdzaan Be'eena Program
- Control (No Intervention): Girls and their female caregivers randomized to the control group will receive 4 retention incentives that are mailed to them monthly. These incentives will each be <$10 per dyad, examples include: water bottles, lanyards, pencil cases and tote bags. The control condition was selected by community members and allows for minimal contamination and/or overlap between the AB curriculum and control group

INTERVENTIONS:
Behavioral: Asdzaan Be'eena Program — The program consists of 11 weekly sessions conducted with girls ages 10-14 and their female caregivers. 5 of the 11 sessions will be taught to groups of 9-13 girls and their female caregivers, and 6 of the sessions will be taught to individual girl/female caregiver dyads. The choice to use a mix of group- and individual sessions is based on findings from the formative phase indicating certain topics should be taught in groups (e.g. Navajo history and reproductive health 101), and certain topics be taught in individual dyads (e.g. family values and the clan system).
  Each of the sessions (group and individual) will be 60-90 minutes in duration and delivered by a trained Family Health Coach (FHC). Group sessions will take place at a local community center in a private room. Individual dyad sessions will take place in the girls'/female caregivers' home or another private place of their choosing, such as our local Johns Hopkins offices.
  Arms: Intervention

SUMMARY:
The objective of this research study is to evaluate a culturally grounded program among American Indian (AI) female adolescents and their female caregivers. Specifically, investigators aim to evaluate the impact of "Asdzaan Be'eena'" or Female Pathways in English (henceforth referred to as AB) on risk and protective factors for early substance use and sexual debut through a randomized controlled trial (RCT) in partnership with the Navajo Nation. The program was developed and pilot tested through an extensive formative phase conducted by our tribal-academic partnership (IRB protocols: #00006569 and #00009117). Investigators will examine the efficacy of the AB program for reducing risk factors and improving protective factors associated with early substance use and sexual debut, with long term goals of reducing teen pregnancy and teen substance use.

DETAILED DESCRIPTION:
American Indian/Alaska Native(AI/AN) communities contend with high rates of poverty and unemployment, as well as historical trauma and adverse events resulting in poor health outcomes and health disparities across their life course. AI youth adolescents are particularly impacted by these health disparities. They are more likely to be sexually active, have their first sexual intercourse at a young age and have higher rates of teen pregnancy and repeat teen pregnancy than other racial/ethnic groups. In 2016, the birth rate for AI/AN teen girls (age 15-19) was 35 per 1,000, well above the national birth rate of 20.3 per 1,000.

Teen pregnancy may lead to lower educational attainment and is associated with a lower annual income for the mother. Nationally, only about 63% of teen mothers obtain a high school diploma and just 2% earn a college degree. Furthermore, studies have found that decades after becoming a parent, teen mothers have lower annual incomes than women who wait to become mothers. The consequences of teen pregnancy continue generations later. Babies born as result of a teen pregnancy are more likely to be premature and of low birth weight, raising their risk for other health problems including blindness, deafness, chronic respiratory problems, mental illness and mental retardation. Children of teen parents are more likely to live in poverty, drop out of high school and themselves become teen parents. The poverty rate for children born to teenage mothers who never married and who did not graduate from high school is 78% (compared to 9% of children born to women over age 20 who are currently married and did graduate from high school).

Compounding teen pregnancy, AI/ANs have the highest substance use and related morbidity and mortality of any U.S. racial group and are more likely to initiate drug and alcohol use before the age of 13. In AI communities, girls and boys have distinct patterns and processes for underage substance use that leads to early initiation of sex and sexual risk-taking. Among AIs, girls are more likely than boys to use substances during adolescence due to poor self-esteem or self-identity. Girls are also more likely than boys to be offered substances in private settings by female relatives. Additionally, poor attachment to parents is a stronger risk factor for substance use among girls than boys. Thus, gender-specific approaches are needed for optimal prevention of adolescent substance use in AI communities.

An intervention that works with AI females together with their female caregivers and incorporates AI cultural strengths and traditions, while also helping girls grow their ethnic identity and self-esteem may prove efficacious in preventing teen pregnancy, reducing early initiation of substance use and progression to misuse, and improving the health and well being of AI girls and families. The Navajo Nation and Johns Hopkins (JHU) have a long-standing history of addressing AI health disparities through culturally tailored and community-engaged programming and are poised to conduct the RCT described herein.

Investigators will evaluate the intervention: "Asdzaan Be'eena: Female Pathways" (AB). The program consists of 11 weekly sessions conducted with girls ages 10-14 and their female caregivers. Five of the 11 sessions will be taught to groups of 9-13 girls and their female caregivers, and 6 of the sessions will be taught to individual girl/female caregiver dyads. The choice to use a mix of group- and individual sessions is based on findings from the formative phase indicating certain topics should be taught in groups (e.g. Navajo history and reproductive health 101), and certain topics be taught in individual dyads (e.g. family values and the clan system).

Each of the sessions (group and individual) will be 60-90 minutes in duration and delivered by a trained Family Health Coach (FHC). Group sessions will take place at a local community center in a private room. Individual dyad sessions will take place in the girls'/female caregivers' home or another private place of their choosing, such as our local Johns Hopkins offices. Transportation to the group sessions will be provided upon request. The program will be conducted over 2.5-3 months with one session occurring every week for 11 weeks. The total program duration is 660-990 minutes. The control condition was selected by community members and allows for minimal contamination and/or overlap between the AB curriculum and control group

ELIGIBILITY:
Inclusion Criteria (Caregivers):

* Female > 18 years of age
* Self-identify as Navajo
* Be a caregiver of a girl 10-14 years old who is available to enroll in the study
* Living within 50 miles of the Chinle, Arizona or Tuba City, Arizona Johns Hopkins program offices
* Willing to complete all assessments
* Willing to be randomized
* Speaks and reads English
* Not cognitively or visually impaired (able to complete assessments)
* Review and sign informed consent

Inclusion Criteria (Youth)

* Female, 10-14 years old
* Have a caregiver enrolled in the study
* Living within 50 miles of the Chinle, Arizona or Tuba City, Arizona Johns Hopkins program offices
* Willing to be randomized
* Willing to complete all assessments
* Speaks and reads English
* Not cognitively or visually impaired (able to complete assessments)
* Review and sign a study assent and have a parent/guardian sign parental permission

Exclusion Criteria:

-

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 408 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Change in youth reported parent-youth communication scale | Baseline, 6- and 12-months post implementation
  Investigators will measure change in youth reported parent-youth communication from baseline and 6- and 12- months post program completion via 9-item communication assessment (5-point Likert scale [0-Never; 4- Everyday). A higher score indicates a better outcome.
Change in parent reported parent-youth communication scale | Baseline, 6- and 12-months post implementation
  Investigators will measure change in parent reported parent-youth communication from baseline and 6- and 12- months post program completion via an 8-item communication assessment (5-point Likert scale [0-Never; 4- Everyday). A higher score indicates a better outcome.
Change in youth reported monitoring | Baseline, 6- and 12-months post implementation
  Investigators will measure change in youth reported monitoring from baseline and 6- and 12- months post program completion via a 5-item parental monitoring assessment (5-point Likert scale [0-Never; 4- Everyday). A higher score indicates a better outcome.
Change in parent reported monitoring | Baseline, 6- and 12-months post implementation
  Investigators will measure change in parent reported monitoring from baseline and 6- and 12- months post program completion via a 9-item parental monitoring assessment (5-point Likert scale [0-Never; 4- Everyday). A higher score indicates a better outcome.
Change in youth reported parental responsiveness | Baseline, 6- and 12-months post implementation
  Investigators will measure change in youth reported parental responsiveness from baseline and 6- and 12- months post program completion via a 5-item authoritative parenting index (4-point Likert scale [0-Not at all like her; 3- Just Like her). A higher score indicates a better outcome.
Change in parent reported parental responsiveness | Baseline, 6- and 12-months post implementation
  Investigators will measure change in parent reported parental responsiveness from baseline and 6- and 12- months post program completion via a 5-item authoritative parenting index (4-point Likert scale [0-Not at all like her; 3- Just Like her). A higher score indicates a better outcome.
Change in proportion of youth who state they plan to delay having sexual intercourse until they graduate from high school | Baseline, 6- and 12-months post implementation
  Change in proportion of youth who report they intend to delay sexual intercourse until they graduate from high school between individuals randomized to the AB program vs. those randomized to the control condition. Proportions will be measured from baseline to 6- and 12-months post program completion via one question. This is completed by the child (0-No; 1-Yes). A higher proportion indicates more youth intend to abstain from sex.
Change in proportion of youth who state they plan to engage in sexual intercourse while they are a teenager | Baseline, 6- and 12-months post implementation
  Investigators will measure change in proportion of youth who report they intend to have sexual intercourse when they are a teenager between individuals randomized to the AB program vs. those randomized to the control condition. Proportions will be measured from baseline to 6- and 12-months post program completion via one question. This is completed by the child (0-No; 1- Yes). A higher proportion indicates more youth intend to have sex when they are a teenager. A higher proportion indicates a worse outcome.
Change in mean score on externalizing and internalizing behaviors | Baseline, 6- and 12-months post implementation
  Investigators will measure change in internalizing and externalizing behaviors between individuals randomized to the AB program vs. those randomized to the control condition. Change in internalizing/externalizing behaviors will be measured via the Achenbach System of Empirically Based Assessment (ASEBA) completed by the caregiver (reporting on child behaviors) (3-point Likert Scale [0-not true; 2-very true]). A higher score across these variables indicates a worse outcome (i.e. higher (more) internalizing and externalizing behaviors).

SECONDARY OUTCOMES:
Change in caregiver parenting self-efficacy | Baseline, 6- and 12-months post implementation
  Investigators will measure change in caregiver parenting self-efficacy from baseline and 6- and 12- months post program completion via a 10-item parenting self-efficacy questionnaire (5-point Likert scale [0-Never; 4-Always]). A higher score indicates a better outcome.
Change in caregiver parenting agency | Baseline and 6- and 12-months post implementation
  Investigators will measure change in caregiver parenting agency from baseline and 6- and 12- months post program completion via a 10-item parenting self-agency questionnaire (5-point Likert scale [0-Never; 4-Always]). A higher score indicates a better outcome.
Change in mean score on healthy relationship skills | Baseline, 6- and 12-months post implementation
  Investigators will measure change in healthy relationship skills between individuals randomized to the AB program vs. those randomized to the control condition. This outcome measures will be assessed from baseline to 6- and 12-months post program completion via the Five Domains of Interpersonal Competence in Peer Relationships, a 7-item questionnaire (0-I'm not good at this; 4-I'm really good at this). A higher score indicates a better outcome.
Change in in youth future aspirations | Baseline, 6- and 12-months post implementation
  Investigators will measure change in youth future aspirations between individuals randomized to the AB program vs. those randomized to the control condition. This outcome measure will be assessed from baseline to 6- and 12-months post-program completion via the Youth Assets Survey (4-point Likert Scale [0-not at all important; 4-somewhat important]). A higher score indicates a better outcome.
Change in youth cultural connectedness | Baseline, 6- and 12-months post implementation
  Change in youth cultural connectedness at 6- and 12-month follow-up between individuals randomized to the AB program vs. those randomized to the control condition. Youth will be assessed on a 7-item scale (4-point Likert Scale [1-strongly disagree; 4-strongly agree]). A higher score indicates a better outcome Time Frame: Baseline, 6- and 12 months post implementation
Change in caregiver cultural connectedness | Baseline and 6- and 12-months post implementation
  Change in caregiver cultural connectedness at 6- and 12-month follow-up between individuals randomized to the AB program vs. those randomized to the control condition. Caregivers will be assessed on an 8-item scale (4-point Likert Scale [1-strongly disagree; 4-strongly agree]). A higher score indicates a better outcome
Change in youth sexual initiation | Baseline, 6- and 12-months post implementation
  Study investigators will compare youth sexual initiation between youth randomized to the AB program vs. those randomized to the control condition. This outcome will be assessed via one question (0-No; 1-Yes). The outcome measure will be reported as a proportion. A higher proportion indicates more youth have had sex.
Change in proportion on youth substance use initiation | Baseline, 6- and 12-months post implementation
  Investigators will measure change in proportion of youth who report they have ever used alcohol, marijuana or other illegal drugs between youth randomized to the AB program vs. those randomized to the control condition. This outcome measure will be assessed from baseline to 6- and 12-months post program completion via one question (0-No; 1- Yes). This is completed by the child. A higher proportion indicates more youth have ever used a substance.
Change in sexual activity, past 3 months | Baseline and 6- and 12-months post implementation
  Change in youth sexual activity, past 3 months at 6 and 12-month follow-up will be compared between individuals randomized to the AB program vs. those randomized to the control condition. This outcome measure will be reported as a proportion. A higher proportion indicates a negative outcome.
Change in youth reported substance use, past 3 months | Baseline and 6- and 12-months post implementation
  Change in youth substance use, past 3 months at 6 and 12-month follow-up, will be compared between individuals randomized to the AB program vs. those randomized to the control condition. This outcome measure will be reported as a proportion. A higher proportion indicates a negative outcome.
Change in family environment and functioning | Baseline and 6- and 12-months post implementation
  Change in family environment and functioning will be compared between youth/caregivers randomized to the AB program vs. those randomized to the control condition. This outcome measure will be assessed using the Family Environment Scale (true=1/false=0). The scale ranges from 0 - 27. A higher score indicates a better outcome.
Change in parental attitudes and expectations related to substance use and sexual intercourse | Baseline and 6- and 12-months post implementation
  Investigators will measure change in parental attitudes and expectations related to substance use and sexual intercourse between those randomized to the AB program vs. those randomized to the control condition. This outcome measure will be assessed from baseline to 6- and 12-months post program completion via a 6-item assessment (5-point Likert scale [0-strongly disagree; 4-strongly agree]) completed by caregivers. A higher score indicates a better outcome.
Change in proportion of caregivers reporting substance use in the past 3 months | Baseline and 6- and 12-months post implementation
  Change in caregiver substance use in the past 3 months at 6- and 12-month follow-up will be compared between individuals randomized to the AB program vs. those randomized to the control condition.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Tingey, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Jennifer Richards, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Center for American Indian Health - Chinle, Chinle, Arizona
  - Center for American Indian Health - Tuba City, Tuba City, Arizona

REFERENCES:
- [Derived] Chambers RA, Begay J, Patel H, Richards J, Nelson D, Rosenstock S, Huskon R, Mitchell K, Begay T, Tingey L. Rigorous evaluation of a substance use and teen pregnancy prevention program for American Indian girls and their female caregivers: a study protocol for a randomized controlled trial. BMC Public Health. 2021 Jun 21;21(1):1179. doi: 10.1186/s12889-021-11131-x. PMID 34154552